CLINICAL TRIAL: NCT00600236
Title: HLA and it Relation With the Development of Proliferative Diabetic Retinopathy in Mexican Population
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: poor accrual
Sponsor: Asociación para Evitar la Ceguera en México (Other)
Collaborators: Instituto Nacional de Referencia Epidemiológica (INdRE) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: APEC-0018
Record Dates: First submitted 2006-06-30; First posted 2008-01-24 (Estimated); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Diabetes Mellitus Type 2; Proliferative Diabetic Retinopathy
Keywords: Diabetes mellitus type 2 with 10 years of diagnosis and no diabetic retinopathy; Diabetes mellitus type 2 with 10 years of diagnosis and proliferative diabetic retinopathy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Blood Specimen Collection

INTERVENTIONS:
Procedure: blood sample

SUMMARY:
One of the first causes of irreversible blindness in mexican population is diabetic retinopathy which is clearly diferent between patients the time of evolution and development of retinopathy and complications. The aim of this study is to explore the inmunogenetic profile and the influence of HLA in this variations of the sickness to predict the severity of diabetic complications.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus type 2 with 10 years of diagnosis and no diabetic retinopathy
* Diabetes mellitus type 2 with 10 years of diagnosis and proliferative retinopathy

Exclusion Criteria:

* Systemic hipertension
* Cardic disease
* Lupus
* Any kind of artritis
* Allergies
* Optic Neuritis
* VKH
* Cancer
* Inmunological diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2004-09; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Quiroz-Mercado, MD, Principal Investigator — Asociación para Evitar la Ceguera en México, Hospital "Luis Sánchez Bulnes"
Locations (1):
- Asociación para Evitar la Ceguera en México, Hospital "Luis Sanchez Bulnes", Mexico City, Mexico DF, Mexico